CLINICAL TRIAL: NCT06819865
Title: EkoSonic Endovascular System in China RWS(ANTEATER)
Brief Title: A Real-World Study of EkoSonic Endovascular System in Chinese Populations With Acute Pulmonary Embolism
Acronym: ANTEATER
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S6364
Record Dates: First submitted 2025-01-15; First posted 2025-02-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Pulmonary Embolism
Keywords: PE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single group observational study: To collect the real-world clinical outcome data of EkoSonicTM Endovascular System in Chinese patients with acute pulmonary embolism during practical clinical care.
  Interventions: Device: EkoSonicTM Endovascular System

INTERVENTIONS:
Device: EkoSonicTM Endovascular System — EkoSonicTM Endovascular System and its upgraded versions if applicable The EkoSonicTM Endovascular System is a non-implanted system comprising a sterile, single-use EkoSonic Endovascular Device (Infusion Catheter and Ultrasonic Core) and reusable EKOSTM Control System 4.0(Control Unit, Connector Interface Cable and power cord).

SUMMARY:
This study to collect the real-world clinical outcome data of EkoSonicTM Endovascular System in Chinese patients with acute pulmonary embolism during practical clinical care.

DETAILED DESCRIPTION:
This is a multi-center, single arm, prospective, observational, real-world study.To collect the real-world clinical outcome data of EkoSonicTM Endovascular System in Chinese patients with acute pulmonary embolism during practical clinical care.

Up to 30 patients will be enrolled in this study and up to 30 patients will be enrolled in this study to observation safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with acute symptomatic pulmonary embolism (Symptomatic duration < 14 days).
2. The right ventricle diameter to left ventricle diameter of end-diastolic dimension ratio ≥1 measured by echocardiographic image
3. Investigator has selected the EkoSonicTM Endovascular System with r-tPA to treat patient.

Exclusion Criteria:

1. The patients with acute symptomatic pulmonary embolism (Symptomatic duration < 14 days).
2. The right ventricle diameter to left ventricle diameter of end-diastolic dimension ratio ≥1 measured by echocardiographic image
3. Investigator has selected the EkoSonicTM Endovascular System with r-tPA to treat patient.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients who received EkoSonicTM Endovascular System treatment with r-tPA for acute pulmonary thromboembolism, and who could provide sufficient echocardiographic quality to assess the collection of primary endpoint, and prospectively collect the clinical data related to the protocol in the actual clinical diagnosis and treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
RV vs LV end-diastolic diameter ratio | after the completion of EKOS treatment 48 hours compared with the baseline
  The change in the right ventricular end-diastolic diameter to left ventricle end-diastolic diameter ratio at 48hours after the completion of EKOS treatment compared with the baseline.

SECONDARY OUTCOMES:
RV vs LV end-diastolic diameter ratio | after the completion of EKOS treatment 24 hours, Discharge(Approximately within 15 days after completed treatment) , after the completion of EKOS treatment Month 1, Month 3, Month 6, compared to the baseline，through study completion, an average of 1 year
  The change in the right ventricle diameter to left ventricle diameter of end-diastolic dimension ratio at 24h, Discharge(Approximately within 15 days after completed treatment) , after the completion of EKOS treatment Month 1, Month 3, Month 6, compared to the baseline.
PE events after the completion of EKOS treatment | After the completion of EKOS treatment 24hours, 48hours,Discharge(Approximately within 15 days after completed treatment), after the completion of EKOS treatment Month 1, Month 3, Month 6, compared to the baseline
  Recurrent symptomatic PE events after the completion of EKOS treatment.
Serious adverse events related to EKOS or procedure | After enrollment to end of study，through study completion, an average of 1 year
  All of SAE related to EKOS or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guangqi Chang, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University